CLINICAL TRIAL: NCT01347125
Title: ImCardia for DHF - Safety and Functionality
Brief Title: ImCardia for DHF to Treat Diastolic Heart Failure (DHF) Patient a Pilot Study
Acronym: ImCardia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: CorAssist believes that certain improvements are needed to the device
Sponsor: CorAssist Cadiovascular Ltd. (Industry)
Responsible Party: Dr. Lea Lak, CorAssist Cardiovascular Ltd.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLD 0201
Record Dates: First submitted 2011-04-28; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: DHF (diastolic heart failure); HFNEF (heart failure with normal ejection fraction
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ImCardia (Experimental): Aortic Stenosis patients candidates for Aortic Valve Replacement (AVR) implanted with the ImCardia device
  Interventions: Device: ImCardia Device
- AVR control group (No Intervention): Aortic stenosis patients candidates for aortic valve replacement

INTERVENTIONS:
Device: ImCardia Device — The device operates by harnessing energy expended by the left ventricle (LV) during Systole and returning it to the heart during Diastole thereby making it available to augment diastolic performance
  Other Names: IMC 01
  Arms: ImCardia

SUMMARY:
This study is designed to evaluate the ImCardia safety and to demonstrate system functionality in patients undergoing AV replacement with respect to 36 months follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female able to understand and sign a informed consent
2. Be 50 years of age or older
3. NYHA class III, IV
4. EF >55%
5. Candidates for aortic valve replacement due to aortic stenosis.
6. Agrees to attend all follow- up evaluations

Exclusion Criteria:

1. Free wall thickness less than11.5mm
2. Adhesions are expected from a previous surgery or medical condition (e.g. s/p chest radiation therapy etc.)
3. Presence of significant myocardial scars (e.g. postinfarction) at proposed site for implant of ImCardia™device Attachment screw.
4. Likely to be need CABG following the implantation of the ImCardia™
5. Intra-cardiac thrombus/mass
6. Myocarditis
7. Acute/chronic pericarditis
8. Not a candidate for sternotomy
9. Active infection
10. Stroke, surgery or ICD within 3 months
11. Acute coronary syndrome during the past 6 months
12. Left ventricular regional wall motion abnormalities
13. Significant valvular disease other that aortic stenosis
14. Significant pulmonary disease
15. A history of alcohol abuse, drug addiction, or other psychosocial condition that would preclude successful participation, or clear judgment and informed consent in the opinion of the Principal Investigator
16. Participating in another trial (other than non-therapeutic or interventional observation) within the last 60 days.
17. History of noncompliance to medical therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Safety: Adverse event reporting | 36 month
  Adverse event reporting will continue up to 36 month follow up. Any complication attributed to the device will be recorded.
  Any Major Adverse Cardiac Event (MACE) will be evaluated in a safety committee composed from company representative and a cardiosurgeon which is not part of the company

SECONDARY OUTCOMES:
Functionality - Successful Device implantation | Immediately post implantation day
  The surgeon will score device implantation procedure post operation.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Lak, M.D., Study Director — CorAssist Cardiovascular